CLINICAL TRIAL: NCT06204107
Title: A Randomized, Open-label, Single Dose, Crossover, Phase Ⅰ Trial to Evaluate the Food Effect on Pharmacokinetic Profiles and Safety of CKD-379 in Healthy Volunteers
Brief Title: A Clinical Trial to Evaluate the Food Effect on Pharmacokinetic Profiles and Safety of CKD-379
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A125_05FDI2310
Record Dates: First submitted 2023-12-17; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): * Phase 1: CKD-379 Test drug
  * Phase 2: CKD-379 Reference drug
  Interventions: Drug: CKD-379(Empagliflozin+sitagliptin+metformin) Test drug; Drug: CKD-379(Empagliflozin+sitagliptin+metformin) Reference drug
- Group 2 (Experimental): * Phase 1: CKD-379 Reference drug
  * Phase 2: CKD-379 Test drug
  Interventions: Drug: CKD-379(Empagliflozin+sitagliptin+metformin) Test drug; Drug: CKD-379(Empagliflozin+sitagliptin+metformin) Reference drug

INTERVENTIONS:
Drug: CKD-379(Empagliflozin+sitagliptin+metformin) Test drug — oral, once
Drug: CKD-379(Empagliflozin+sitagliptin+metformin) Reference drug — oral, once

SUMMARY:
This is a randomized, open-label, single dose, crossover, phase Ⅰ trial to evaluate the food effect on pharmacokinetic profiles and safety of CKD-379 in healthy volunteers

DETAILED DESCRIPTION:
Participants were randomly assigned in a 1:1 ratio. The patients are prescribed oral administration of the appropriate IP(2 tablets in single dose: actual medication)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 54 years
* BMI measurement result is 18.0 kg/m2 to 30 kg/m2
* Written informed consent
* Other inclusion criteria, as defined in the protocol

Exclusion Criteria:

* History of clinically significant liver, kidney, blood, digestive, respiratory, endocrine, cardiovascular, neurological, mental, or immune system disorders
* AST or ALT or total bilirubin > 1.5 times the upper limit of normal range
* History of regular alcohol consumption > 21 units/week within 6 months at the time of screening
* Participated in a clinical trial within 6 months prior to 1st IP dosing
* Other exclusive inclusion criteria, as defined in the protocol

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
AUCt of Empagliflozin, sitagliptin, metformin | 0 hour ~ 48 hour after drug administration
Cmax of Empagliflozin, sitagliptin, metformin | 0 hour ~ 48 hour after drug administration

SECONDARY OUTCOMES:
AUCinf of Empagliflozin, sitagliptin, metformin | 0 hour ~ 48 hour after drug administration
Tmax of Empagliflozin, sitagliptin, metformin | 0 hour ~ 48 hour after drug administration
t1/2 of Empagliflozin, sitagliptin, metformin | 0 hour ~ 48 hour after drug administration
CL/F of Empagliflozin, sitagliptin, metformin | 0 hour ~ 48 hour after drug administration
Vd/F of Empagliflozin, sitagliptin, metformin | 0 hour ~ 48 hour after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyong Jeong, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No